CLINICAL TRIAL: NCT00989963
Title: A 12-week, Double-blind, International, Multicenter, Dose-response Study of the Safety and Efficacy of Beraprost Sodium Modified Release (BPS-MR) in Patients With Pulmonary Arterial Hypertension (PAH)
Brief Title: Dose-response Study of the Safety and Efficacy of Beraprost Sodium Modified Release (BPS-MR) in Patients With Pulmonary Arterial Hypertension (PAH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lung Biotechnology PBC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BPS-MR-PAH-203
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Results first posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Maximum Tolerated Dose (MTD) (Experimental): Patients in the MTD treatment group will dose escalate weekly by 60µg b.i.d. until they reach the maximum dose of 600µg b.i.d. or they reach an intolerable dose which requires them to down-titrate by 60µg b.i.d. In these instances and at the Investigator's discretion, further attempts at dose escalation may be made.
  Interventions: Drug: Beraprost Sodium Modified Release
- Low Fixed Dose (Experimental): The low dose group will receive 60µg twice a day(b.i.d.)
  Interventions: Drug: Beraprost Sodium Modified Release
- High Fixed Dose (Experimental): Patients in the high dose group will dose escalate weekly by 60µg twice a day (b.i.d.) until they reach the fixed dose of 240µg b.i.d. Once patients in these treatment groups have reached their assigned maximum dose of active drug,
  Interventions: Drug: Beraprost Sodium Modified Release

INTERVENTIONS:
Drug: Beraprost Sodium Modified Release — 60µg Tablets, twice a day for 12 weeks

SUMMARY:
This is a 12-week, international, multicenter, double-blind, three-group, dose-response study to assess the safety and efficacy of BPS-MR in patients with PAH. Eligible patients will have been previously diagnosed with PAH and will be on a stable course of an ERA and/or PDE-5 inhibitor for at least 60 days prior to Baseline.

Patients will be randomized to 1 of 3 treatment groups in a 1:1:1 ratio and will be stratified by PAH background therapy (Endothelium Receptor Antagonist (ERA), Phosphodiesterase-5 (PDE-5), and both). The treatment groups consist of one Maximum Tolerated Dose (MTD) and two Fixed Dose (FD) groups. Following randomization, patients will begin taking active drug (60µg) orally twice daily. Patients will visit their investigational site at Week 6 and Week 12 for study evaluations.

DETAILED DESCRIPTION:
This is a 12-week, international, multicenter, double-blind, three-group, dose-response study to assess the safety and efficacy of BPS-MR in patients with PAH. Eligible patients will have been previously diagnosed with PAH and will be on a stable course of an ERA and/or PDE-5 inhibitor for at least 60 days prior to Baseline.

A total of approximately 36 patients will be randomized to 1 of 3 treatment groups (12 per group) in a 1:1:1 ratio and will be stratified by PAH background therapy (ERA, PDE-5, and both). The treatment groups consist of one MTD and two FD groups. Following randomization, patients will begin taking active drug (60µg) orally twice daily. Patients will visit their investigational site at Week 6 and Week 12 for study evaluations. Between visits, clinical site personnel will contact patients by phone each week to assess tolerability, provide instructions for a change in dosage, record changes in concomitant medications, and record adverse events. Patients who complete the study will be offered the opportunity to continue taking study medication in a separate open-label continuation protocol. Patients who withdraw early from the study or who otherwise do not elect to enroll into the open-label continuation protocol will be down-titrated off of BPS-MR at the discretion of the Investigator, at a maximum decrement not to exceed one tablet (60µg) b.i.d. per day and a minimum decrement of one tablet (60µg) b.i.d. per week.

Patients in the iMTD treatment group will dose escalate weekly by 60µg b.i.d. until they reach the maximum dose of 600µg b.i.d. or they reach an intolerable dose which requires them to down-titrate by 60µg b.i.d. In these instances and at the Investigator's discretion, further attempts at dose escalation may be made.

The FD treatment groups will consist of a low dose group receiving 60µg b.i.d. and a high dose group receiving 240µg b.i.d. Patients in the high dose group will dose escalate weekly by 60µg b.i.d. until they reach the fixed dose of 240µg b.i.d. Once patients in these treatment groups have reached their assigned maximum dose of active drug, weekly increases in the number of placebo tablets administered will continue in order to maintain the blind.

Patients will be requested to maintain a daily diary of symptoms and study drug administration for evaluation by clinical site personnel. Also, patients will be given the option to contribute blood for pharmacokinetic assessment of BPS/BPS-314d plasma concentrations at the Week 12 visit.

ELIGIBILITY:
Inclusion Criteria:

1. IRB approved written informed consent has been obtained.
2. Male or female, age 18 to 75 years (inclusive).
3. Established diagnosis of pulmonary arterial hypertension that is either idiopathic or familial PAH, collagen vascular disease associated PAH, PAH induced by anorexigens, or PAH associated with repaired congenital systemic-to-pulmonary shunts (repaired ≥5 years).
4. Clinically stable PAH as determined by the Investigator.
5. Able to walk unassisted.
6. Has a complete, unencouraged 6MWT distance of 150 to 450 meters (inclusive) at Screening.
7. Previous (at any time) right heart cardiac catheterization with findings consistent with PAH, specifically mean Pulmonary Arterial Pressure (PAPm) ≥25 mmHg (at rest), Pulmonary Capillary Wedge Pressure (PCWP) (or left ventricular end diastolic pressure) ≤15 mmHg, and Pulmonary Vascular Resistance (PVR) >3 mmHg/L/min.
8. Previous (at any time) chest radiograph consistent with the diagnosis of PAH.
9. Has been on a stable course of an ERA or/and PDE-5 inhibitor for a minimum of 60 days prior to Baseline.
10. Women of child-bearing potential (defined as less than 1 year post-menopausal or not surgically sterile) must be using an acceptable method of birth control or practicing abstinence. If sexually active, female patients must use a double barrier method of birth control, such as a condom and spermicidal. Patient must have a negative pregnancy test at the Screening and Baseline visits.
11. Willing and able to comply with study requirements and restrictions.

Exclusion Criteria:

1. Has pulmonary venous hypertension, pulmonary veno-occlusive disease, pulmonary capillary hemangiomatosis, or chronic thromboembolic pulmonary hypertension.
2. Has a history of interstitial lung disease, unless:

   * Pulmonary Function Testing conducted within 6 months of the Baseline visit demonstrates a Total Lung Capacity ≥ 70 % of predicted.
3. Has a history of obstructive lung disease, unless:

   * Pulmonary Function Testing conducted within 6 months of the Baseline visit demonstrates a forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) ratio of ≥ 50%.
4. Is pregnant and/or lactating.
5. Changed or discontinued any PAH medication within 60 days prior to the Baseline visit including, but not limited to, an ERA, PDE-5 inhibitor, or calcium channel blocker (with the exception of anticoagulants).
6. Has an ongoing hemorrhagic condition (e.g. upper digestive tract hemorrhage, hemoptysis, etc), or has a pre-existing condition that, in the Investigator's judgment may increase the risk for developing hemorrhage during the study (e.g. hemophilia). Transient hemorrhage (e.g. epistaxis, normal menstrual bleeding, gingival bleeding, hemorrhoidal hemorrhage, etc.) will not preclude enrollment.
7. Has donated blood or plasma, or has lost a volume of blood >450mL within 6-weeks of the Baseline visit.
8. Has received any investigational medication, device or therapy within 30 days prior to the Baseline visit or is scheduled to receive another investigational drug, device or therapy during the course of the study.
9. Has received any prostanoid therapy at any time.
10. Has any preexisting disease known to cause pulmonary hypertension other than collagen vascular disease.
11. Has any musculoskeletal disease or any other disease that would limit ambulation.
12. Has any form of unrepaired or recently repaired (< 5 years) congenital systemic-to-pulmonary shunt other than patent foramen ovale.
13. History of pulmonary embolism or deep venous thrombosis.
14. History of ischemic heart disease, including previous myocardial infarction, or symptomatic coronary artery disease, or history of left sided myocardial disease as evidenced by a mean PCWP (or a left ventricular end diastolic pressure) > 15 mmHg or left ventricular ejection fraction < 40% as assessed by either multigated angiogram, angiography or echocardiography, or left ventricular shortening fraction < 22% as assessed by echocardiography. Note that patients in whom abnormal left ventricular function is attributed entirely to impaired left ventricular filling due to the effects of right ventricular overload (i.e. right ventricular hypertrophy and/or dilatation) will not be excluded.
15. Presence of atrial fibrillation (determined from 12-lead ECG at Screening).
16. Any other clinically significant illness that, in the opinion of the Investigator, might put the patient at risk of harm during the study or might adversely affect the interpretation of the study data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2011-09-13 (Actual); Study Completion 2011-09-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (6):
  - Harbor-UCLA Medical Center, Torrance, California
  - Edward Heart Hospital, Naperville, Illinois
  - Beth Israel Medical Center, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
- Belgium (2):
  - Universite Libre de Bruxelles, Bruxellas
  - Catholic University of Leuven, Leuven
- General Teaching Hospital, Prague, Czechia
- Germany (4):
  - Klinikum der Universitat zu Koln, Cologne
  - Medizinische Klinik und Poliklinik, Dresden
  - Abt. Innere Medizin III, Medizinische Universitatsklinik, Heidelberg
  - Universitatsklinik Leipzig Abteilung Pulmologie, Leipzig
- Mater Misericordiae University Hospital Ltd., Dublin, Ireland
- Romania (3):
  - Institutul de Urgenta pentru Boli, Bucharest
  - Institutul National de Pneumologie, Bucharest
  - Institutul de Boli Cardiovasculare, Lasi

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Fixed Dose Group (60 ug): Participants in the low dose group received 60 microgram of Beraprost sodium modified release tablets, orally twice daily up to maximum duration of Week 12.
- High Fixed Dose (FD) Group (240 ug): Participants in the high dose group received starting dose of 60 microgram of Beraprost sodium modified release tablets twice daily which was escalated until they reached the fixed maximum dose of 240 microgram twice daily up to a maximum duration of Week 12
- Maximum Tolerated Dose (MTD): Participants in this group received starting dose of 60 microgram of Beraprost sodium modified release tablets twice daily which was escalated until they reached the fixed maximum dose of 600 microgram twice daily up to a maximum duration of Week 12 or they reached an intolerable dose which required them to down-titrate by 60 microgram twice daily in these instances and at the Investigator's discretion, further attempts at dose escalation may have been made.
Period: Overall Study
Arm/Group | Low Fixed Dose Group (60 ug) | High Fixed Dose (FD) Group (240 ug) | Maximum Tolerated Dose (MTD)
Started (Full Analysis Population: All randomized participants (per intended treatment assignment).) | 12 | 12 | 12
Safety Population (Randomized participants (per actual treatment received) who received ≥1 dose of study drug.) | 13 (1 participant randomized to MTD received FD 60 ug; was included in FD 60 ug arm for this population) | 12 | 11 (1 participant randomized to MTD received FD 60 ug; was included in FD 60 ug arm for this population)
Per-Protocol Population (Randomized participants (actual treatment received), completed study, no major protocol deviations.) | 12 (1 participant randomized to MTD received FD 60 ug; was included in FD 60 ug arm for this population) | 11 | 10 (1 participant randomized to MTD received FD 60 ug; was included in FD 60 ug arm for this population)
Completed | 11 | 11 | 11
Not Completed | 1 | 1 | 1
Not completed — Adverse Event | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who were randomized in the study (per intended treatment assignment).
Groups:
- High Fixed Dose Group (240 ug): Participants in the high dose group received starting dose of 60 microgram of Beraprost sodium modified release tablets twice daily which was escalated until they reached the fixed maximum dose of 240 microgram twice daily up to a maximum duration of Week 12
- Total: Total of all reporting groups
Arm/Group | Low Fixed Dose Group (60 ug) | High Fixed Dose Group (240 ug) | Maximum Tolerated Dose (MTD) | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (14.19) | 45.1 (15.2) | 51.1 (14.71) | 47.4 (14.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 30
  Male | 2 | 2 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 4 | 6
  Not Hispanic or Latino | 12 | 10 | 8 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 12 | 11 | 12 | 35
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Pulmonary Vascular Resistance (PVR) [Mean (Standard Deviation); unit: Wood Units (mmHg/L/min)] — Pulmonary Vascular Resistance the difference between is the mean pulmonary arterial pressure and the left atrial filling pressure divided by the cardiac output. Population: Randomized participants (actual treatment received) who had completed the study and had received the required protocol processing for the study, i.e., no major protocol deviations (Per-Protocol Population).
  Wood Units (mmHg/L/min)
    number analyzed (Participants) | 12 | 11 | 10 | 33
    (all) | 9.74 (5.35) | 9.39 (4.05) | 10.19 (5.61) | 9.76 (4.89)
Cardiac Output (CO) [Mean (Standard Deviation); unit: Liters per minute (L/min)] — Cardiac Output is the effective volume of blood expelled by either ventricle of the heart per unit of time (generally per minute); it usually refers to left ventricle output. It is equal to the stroke volume multiplied by the heart rate. Population: Randomized participants (actual treatment received) who had completed the study and had received the required protocol processing for the study, i.e., no major protocol deviations (Per-Protocol Population).
  Liters per minute (L/min)
    number analyzed (Participants) | 12 | 11 | 10 | 33
    (all) | 4.44 (1.12) | 5.53 (1.79) | 4.52 (1.20) | 4.83 (1.45)
Mean Pulmonary Arterial Pressure (mPAP) [Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)] — Mean Pulmonary Arterial Pressure (mPAP) is a directly measured hemodynamic parameter. mPAP is recorded during right heart catheterization. Population: Randomized participants (actual treatment received) who had completed the study and had received the required protocol processing for the study, i.e., no major protocol deviations (Per-Protocol Population).
  Millimeters of Mercury (mmHg)
    number analyzed (Participants) | 12 | 11 | 10 | 33
    (all) | 49.58 (18.72) | 57.91 (19.03) | 52.40 (15.54) | 53.21 (17.73)
Six Minute Walk Distance [Mean (Standard Deviation); unit: meters (m)] — Population: Randomized participants (actual treatment received) who had completed the study and had received the required protocol processing for the study, i.e., no major protocol deviations (Per-Protocol Population).
  meters (m)
    number analyzed (Participants) | 12 | 11 | 10 | 33
    (all) | 362.92 (51.01) | 388.73 (74.21) | 327.70 (94.48) | 360.85 (75.75)
Borg Dyspnea Score [Mean (Standard Deviation); unit: scores on a scale] — Population: Randomized participants (actual treatment received) who had completed the study and had received the required protocol processing for the study, i.e., no major protocol deviations (Per-Protocol Population).
  scores on a scale
    number analyzed (Participants) | 12 | 11 | 10 | 33
    (all) | 2.71 (1.48) | 3.36 (2.34) | 3.10 (2.27) | 3.05 (2.00)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pulmonary Vascular Resistance at Week 12
Description: The change in Pulmonary Vascular Resistance (PVR) was evaluated from Baseline to Week 12. PVR is expressed in Wood Units or millimeters of Mercury per Liter per minute (mmHG/L/min)
Time Frame: Week 12
Population: Randomized participants (actual treatment received) who had completed the study and had received the required protocol processing for the study, i.e., no major protocol deviations (Per-Protocol Population).
Measure: Mean (Standard Deviation); unit: Wood Units (mmHg/L/min)
Arm/Group | Low Fixed Dose Group (60 ug) | High Fixed Dose Group (240 ug) | Maximum Tolerated Dose (MTD)
Number analyzed (Participants) | 12 | 11 | 10
Wood Units (mmHg/L/min) | 0.37 (3.08) | 0.00 (1.57) | 0.13 (3.21)

2. Primary Outcome: Change From Baseline in Cardiac Output (CO) at Week 12
Description: The change in Cardiac Output was evaluated from Baseline to Week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters per minute (L/min)
Arm/Group | Low Fixed Dose Group (60 ug) | High Fixed Dose Group (240 ug) | Maximum Tolerated Dose (MTD)
Number analyzed (Participants) | 12 | 11 | 10
Liters per minute (L/min) | 0.16 (1.17) | 0.07 (0.84) | 0.35 (1.15)

3. Primary Outcome: Change From Baseline in Pulmonary Arterial Pressure at Week 12
Description: The change in mean Pulmonary Arterial Pressure (mPAP) was evaluated from Baseline to Week 12.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Low Fixed Dose Group (60 ug) | High Fixed Dose Group (240 ug) | Maximum Tolerated Dose (MTD)
Number analyzed (Participants) | 12 | 11 | 10
mmHg | 0.42 (5.76) | -1.45 (11.96) | 4.10 (5.15)

4. Secondary Outcome: Change in Six Minute Walk Distance From Baseline to Week 6 and Week 12
Description: Area used for the Six Minute Walk Test (6MWT) was pre-measured at 30 meters in length. Rest periods were allowed if patient could no longer continue. If patient needed to rest, he/she could stand or sit and then begin again when rested but the clock continued to run. At the end of 6 minutes, the tester called "stop" while stopping the watch and then measured the distance walked. For purposes of the 6MWT, if patient was assessed at Baseline using oxygen therapy, all future 6MWT were conducted in the same manner. All efficacy results are descriptive; no statistical analysis was conducted.
Time Frame: Baseline, Week 6 and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Low Fixed Dose Group (60 ug) | High Fixed Dose Group (240 ug) | Maximum Tolerated Dose (MTD)
Number analyzed (Participants) | 12 | 11 | 10
meters
  Week 6 Peak | 2.17 (112.63) | 29.91 (46.83) | 39.90 (47.59)
  Week 12 Peak: number analyzed (Participants) | 11 | 11 | 10
  Week 12 Peak | 52.82 (70.53) | 42.18 (83.08) | 47.10 (48.39)
  Week 12 Trough: number analyzed (Participants) | 10 | 9 | 9
  Week 12 Trough | 44.00 (50.74) | 47.67 (92.20) | 11.67 (72.25)

5. Secondary Outcome: Number of Participants in Each World Health Organization (WHO) Functional Class for Pulmonary Arterial Hypertension (PAH) at Week 6 and 12
Description: WHO functional classification for PAH range from Class I (no limitation in physical activity, no dyspnea with normal activity), Class II (slight limitation of physical activity), Class III (marked limitation of physical activity) and Class IV (cannot perform a physical activity without any symptoms, dyspnea at rest).
Time Frame: Week 6 and Week 12
Population: Randomized participants (actual treatment received) who had completed the study and had received the required protocol processing for the study, i.e., no major protocol deviations (Per-Protocol Population). Here, number analyzed signifies number of participants evaluable at specified time points only.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Fixed Dose Group (60 ug) | High Fixed Dose Group (240 ug) | Maximum Tolerated Dose (MTD)
Number analyzed (Participants) | 12 | 11 | 10
Participants
  Week 6: Class I | 1 | 0 | 0
  Week 6: Class II | 6 | 3 | 3
  Week 6: Class III | 5 | 8 | 7
  Week 6: Class IV | 0 | 0 | 0
  Week 12: Class I | 1 | 1 | 0
  Week 12: Class II | 5 | 4 | 3
  Week 12: Class III | 6 | 6 | 7
  Week 12: Class IV | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With at Least One Post-baseline Clinically Significant Laboratory Value
Description: Post-baseline clinically significant values, as defined by the Investigator, for hematology, serum chemistry, coagulation and urinalysis parameters were summarized.
Time Frame: Up to Week 12
Population: Randomized participants (per actual treatment received) who received ≥1 dose of study drug (Safety Population). Overall number of participants analyzed signifies those who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Low Fixed Dose Group (60 ug) | High Fixed Dose Group (240 ug) | Maximum Tolerated Dose (MTD)
Number analyzed (Participants) | 12 | 11 | 11
participants | 5 | 3 | 3

7. Secondary Outcome: Number of Participants With Newly Occurring Clinically Significant ECG Abnormalities
Description: Clinically significant ECG abnormalities at Baseline only are excluded.
Time Frame: Up to 12 weeks
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Low Fixed Dose Group (60 ug) | High Fixed Dose Group (240 ug) | Maximum Tolerated Dose (MTD)
Number analyzed (Participants) | 13 | 12 | 11
Participants
  Right Atrial Abnormality | 0 | 2 | 0
  Chronic Pulmonary Disease Pattern | 0 | 1 | 0
  Low QRS Voltage | 0 | 0 | 1
  Non-Specific ST-T Changes | 0 | 0 | 1

8. Secondary Outcome: Change in Borg Dyspnea Score From Baseline to Week 6 and Week 12
Description: The modified 0-10 category-ratio Borg scale consists of an 11-point scale rating the maximum level of dyspnea experienced during the 6MWT. Scores range from 0 (for the best condition) and 10 (for the worst condition) with nonlinear spacing of verbal descriptors of severity corresponding to specific numbers. The participant chose the number or the verbal descriptor to reflect presumed ratio properties of sensation or symptom intensity. Only participants with both a measurement at baseline and at the given visit are presented. All efficacy results are descriptive; no statistical analysis was conducted.
Time Frame: Baseline, Week 6 and 12
Population: Randomized participants (actual treatment received) who had completed the study and had received the required protocol processing for the study, i.e., no major protocol deviations (Per-Protocol [PP] Population).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Low Fixed Dose Group (60 ug) | High Fixed Dose Group (240 ug) | Maximum Tolerated Dose (MTD)
Number analyzed (Participants) | 12 | 11 | 10
scores on a scale
  Week 6 | 0.71 (1.29) | 0.68 (1.65) | 0.80 (3.13)
  Week 12 at peak: number analyzed (Participants) | 11 | 11 | 10
  Week 12 at peak | 0.50 (0.81) | 0.64 (2.16) | 0.40 (2.69)
  Week 12 at trough: number analyzed (Participants) | 10 | 9 | 9
  Week 12 at trough | 0.45 (0.83) | 1.11 (0.78) | 0.67 (3.00)

9. Secondary Outcome: N-Terminal ProB-type Natriuretic Peptide Level at Week 6 and Week 12
Description: NT-proBNP functions as a strong indicator of prognosis in patients with pulmonary arterial hypertension.
Time Frame: Week 6 and Week 12
Population: Randomized participants (actual treatment received) who completed the study and received required protocol processing, ie, no major protocol deviations (PP Population). Overall number of participants analyzed signifies those who were evaluable for the outcome measure; number analyzed signifies those who were evaluable at specified timepoint only.
Measure: Mean (Standard Deviation); unit: nanograms per Liter (ng/L)
Arm/Group | Low Fixed Dose Group (60 ug) | High Fixed Dose Group (240 ug) | Maximum Tolerated Dose (MTD)
Number analyzed (Participants) | 11 | 10 | 10
nanograms per Liter (ng/L)
  Week 6 | 6.38 (1.28) | 5.82 (0.72) | 6.83 (1.18)
  Week 12: number analyzed (Participants) | 11 | 10 | 9
  Week 12 | 6.33 (1.41) | 6.06 (1.08) | 6.85 (1.55)

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after last dose of study drug (up to Week 12).
Description: Randomized participants (per actual treatment received) who received ≥1 dose of study drug (Safety Population).
Arm/Group | Low Fixed Dose Group (60 ug) | High Fixed Dose Group (240 ug) | Maximum Tolerated Dose (MTD)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 3/13 | 0/12 | 1/11
Other Adverse Events (participants affected / at risk) | 13/13 | 11/12 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Fixed Dose Group (60 ug) (N=13) | High Fixed Dose Group (240 ug) (N=12) | Maximum Tolerated Dose (MTD) (N=11)
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Fixed Dose Group (60 ug) (N=13) | High Fixed Dose Group (240 ug) (N=12) | Maximum Tolerated Dose (MTD) (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 2 | 1 | 4
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 1
Myodesopsia (Eye disorders) | 1 | 0 | 0
Retinal artery occlusion (Eye disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 3 | 7
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 4
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Breath odour (Gastrointestinal disorders) | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 2
Pain (General disorders) | 1 | 1 | 2
Chest discomfort (General disorders) | 2 | 0 | 1
Chest pain (General disorders) | 1 | 1 | 1
Oedema peripheral (General disorders) | 2 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 2
Blood pressure decreased (Investigations) | 1 | 0 | 0
N-terminal prohormone brain natriuretic peptide (Investigations) | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 3
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 6 | 8 | 9
Dizziness (Nervous system disorders) | 2 | 4 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1
Mood swings (Psychiatric disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Polymenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 2 | 4
Hot flush (Vascular disorders) | 1 | 3 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Pallor (Vascular disorders) | 1 | 0 | 0
Vein disorder (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days